CLINICAL TRIAL: NCT00569556
Title: Effect of Care Management on Diabetes Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Areef Ishani, MD, MS, Minneapolis VAMC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3823-A; VISN23
Record Dates: First submitted 2007-12-05; First posted 2007-12-07 (Estimated); Last update posted 2009-06-15 (Estimated); Status verified 2009-06

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Chronic Care Model; Case Management
MeSH Terms: conditions — Diabetes Mellitus | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Patients receive care through primary care provider
  Interventions: Other: Case Management
- Case Management (Experimental): Specially trained nurse case managers contact patients by telephone; monitor blood pressure, LDL, and HgbA1C;, and recommend lifestyle and medication changes as needed
  Interventions: Other: Case Management

INTERVENTIONS:
Other: Case Management — Phone contact by specially trained nurse case managers; lifestyle recommendations and medication changes as needed

SUMMARY:
The purpose of the study is to determine if a nurse managed, protocol driven, disease management process for diabetes results in improved attainment of therapeutic goals for diabetes compared to usual care. It is hypothesized that implementation of the disease management process will improve the percentage of diabetic individuals attaining all three therapeutic targets (HgbA1C<8.0%, LDL<100mg/dl, and BP<130/80mmHG) by 10% compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled at Minneapolis VAMC
* Type 1 or 2 diabetes
* Blood pressure at screening visit > 140mmHg systolic or > 90mmHg diastolic OR HgbA1C at screening visit > 9.0% OR LDL at screening visit > 100mg/dL

Exclusion Criteria:

* Primary care provider unwilling to have participant included in study
* Life expectancy < 1 year
* Unable to give consent
* Severe mental health condition
* pregnant or planning on becoming pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Combined outcome of BP<130/80 mmHG, HgbA1C<8%, and LDL<100mg/dl at 1 year; the primary analysis will compare the intervention to usual care with respect to the percentage of diabetic individuals achieving all three therapeutic goals | one year

SECONDARY OUTCOMES:
Safety of the intervention (occurence of adverse events over the course of the trial) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Areef Ishani, MD, MS, Principal Investigator — Minneapolis VAMC; Nacide Ercan-Fang, MD, Principal Investigator — Minneapolis VAMC
Locations (1):
- Minneapolis Veterans Affairs Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Ishani A, Greer N, Taylor BC, Kubes L, Cole P, Atwood M, Clothier B, Ercan-Fang N. Effect of nurse case management compared with usual care on controlling cardiovascular risk factors in patients with diabetes: a randomized controlled trial. Diabetes Care. 2011 Aug;34(8):1689-94. doi: 10.2337/dc10-2121. Epub 2011 Jun 2. PMID 21636796